CLINICAL TRIAL: NCT01487694
Title: Cimicifuga Racemosa Rhizome and Root Extract for the Management of Moderate to Severe Menopausal Symptoms in Thai Women: a Randomized Controlled Trial
Brief Title: Black Cohosh Extract for the Management of Moderate to Severe Menopausal Symptoms in Thai Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si573/2011
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Hot Flashes
Keywords: back cohosh; cimicifuga racemosa; menopausal symptoms; hot flashes; Kupperman index; MENQOL
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cimicifuga racemosa (Experimental): patients receive cimicifuga racemosa rhizome and root extract 40 mg/day (equivalent to triterpene glycosides 12.3 mg)
  Interventions: Drug: cimicifuga racemosa
- Placebo (Placebo Comparator): Placebo containing no active ingredient which match the drug in bottle, shape, color and smell
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cimicifuga racemosa — Cimicifuga racemosa (black cohosh) rhizome and root extract 40 mg once daily for 12 weeks (equivalent to triterpene glycosides 12.3 mg)
  Arms: Cimicifuga racemosa
Drug: placebo — matching placebo without active ingredient 1 tab daily for 12 weeks
  Arms: Placebo

SUMMARY:
Cimicifuga racemosa (black cohosh) rhizome and root extract have been used to treat menopausal symptoms. To date, there are still scarce information about its efficacy in Thai women with menopausal symptoms. The purpose of this study will assess the efficacy of black cohosh extract in management of menopausal symptoms in Thai women.

ELIGIBILITY:
Inclusion Criteria:

* Thai women, aged ≥ 40 years
* Peri- or postmenopause
* Moderate to severe menopausal symptoms from Kupperman menopausal index score at least 20

Exclusion Criteria:

* Using any drugs or hormonal treatment within 1 month before enrollment
* BMI ≥ 30 kg/m2
* Allergic to drugs or any ingredient
* Liver disease or AST ≥ 37 U/L or ALT ≥ 40 U/L or total bilirubin ≥ 1 mg/dL or direct bilirubin ≥ 0.3 mg/dL
* Psychiatric disease
* Alcohol consumption or any elicit drug use
* Vegetarian (may consume more phytoestrogen)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Mean differences of Kupperman index | 12 weeks

SECONDARY OUTCOMES:
Frequencies of menopausal symptoms | 12 weeks
Compliance | 12 weeks
adverse events | 12 weeks
Mean differences of liver function test | 12 weeks
quality of life | 12 weeks
  Thai MENQOL measurement
Overall satisfaction | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patsama Vichinsartvichai, MD, Principal Investigator — Gynecologic Endocrinology Unit, Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Gynecologic Endocrinology Unit, Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand